CLINICAL TRIAL: NCT02913365
Title: Etiologies, Investigations and Outcomes of Patients Presenting With Hemoptysis in a North-American Tertiary Center at the Beginning of the 21st Century
Brief Title: Etiologies, Investigations and Outcomes of Patients Presenting With Hemoptysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Brian Grondin-Beaudoin, Medical Doctor, Université de Sherbrooke
Other Study IDs: 12-099
Record Dates: First submitted 2016-09-15; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Hemoptysis; Haemoptysis; Lung Disease; Pneumonia; Tuberculosis; Bronchiectasis; Respiratory Tract Infections; Respiratory Tract Diseases; Bronchitis; Mycobacterium Infections; Bronchial Disease; Pulmonary Hemorrhage; Signs and Symptoms; Signs and Symptoms, Respiratory; Pathologic Processes; Mycosis; Hemorrhage; Lung Cancer; Pulmonary Embolism; Arteriovenous Fistula
Keywords: Haemoptysis; Hemoptysis; Airway bleeding; Pulmonary hemorrhage
MeSH Terms: conditions — Hemoptysis; Lung Diseases; Pneumonia; Tuberculosis; Bronchiectasis; Respiratory Tract Infections; Respiratory Tract Diseases; Bronchitis; Mycobacterium Infections; Bronchial Diseases; Signs and Symptoms; Signs and Symptoms, Respiratory; Pathologic Processes; Mycoses; Hemorrhage; Lung Neoplasms; Pulmonary Embolism; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients presenting with hemoptysis: Patients over 18 years of age presenting with hemoptysis at the Centre Hospitalier Universitaire de Sherbrooke (CHUS) between the periods of 2005 to 2010.

SUMMARY:
The study consist of a retrospective analysis of the etiologies, investigations and outcomes of patients presenting between 2005 to 2010 with hemoptysis in a North-American Tertiary center.

DETAILED DESCRIPTION:
RATIONALE:

Hemoptysis, mild or massive, is worrisome for both patients and physicians. The management is different depending on the causes, which are not well defined for the North American population. Despite the fact that this symptom is commonly reported in clinic, there are only a few studies published on this subject in the North-American population. Tuberculosis was a frequent cause of hemoptysis described in populations overseas, which seems less prevalent in the investigators center.

Also, there are no known official guidelines regarding the investigation and management of hemoptysis. The investigators hypothesized that the use of modern technology in a North American population may result in different findings and provide a more accurate diagnostic approach.

Therefore, the study compares the different etiologies of hemoptysis and investigation modalities used in patients presenting in a North-American tertiary center.

METHOD:

The investigators did a retrospective analysis of medical chart from patients with hemoptysis who visited the investigators center between 2005 and 2010. Each visit has been reviewed individually to describe the characteristics of patients, etiologies of hemoptysis and investigation modalities used. All-cause mortality at 2 years was also recorded.

Descriptive statistical analyses will conducted on the data available.

ELIGIBILITY:
Inclusion Criteria:

Any patient over the age of 18 presenting with:

* A diagnosis of hemoptysis on an outpatient basis.
* A diagnosis of hemoptysis during consultation in the emergency department.
* A diagnosis of hemoptysis on the admission sheet.
* A diagnosis of hemoptysis when hospitalized.
* A complication of hemoptysis
* Hemoptysis on the report of the bronchoscopy, chest computed tomography, pulmonary angiography, ventilation-perfusion single-photon emission computed tomography or blood transfusion.

Exclusion Criteria:

* Patients under 18 years of age.
* Patient who refused investigation for hemoptysis.
* Incomplete medical chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient presenting with hemoptysis at the Centre Hospitalier Universitaire de Sherbrooke on an outpatient basis, emergency department or hospitalized at hopital Fleurimont or Hotel-Dieu of Sherbrooke.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Etiologies of hemoptysis | 5 years
  Defining the prevalence of pulmonary diseases by measuring the percentage of patients presenting with hemoptysis caused by lung cancer, bronchiectasis, pulmonary embolism, arteriovenous fistula, pneumonia, bronchitis, tuberculosis, mycosis, heart failure, pseudohemoptysis, cryptogenic and other causes.

SECONDARY OUTCOMES:
Sensitivity of chest X-ray, chest CT-scan and CT-angiography, bronchoscopy, ventilation-perfusion with single-photon emission computed tomography and pulmonary angiography. | 5 years
  Determining the sensitivity in obtaining the etiology of the hemoptysis episode of each diagnostic modality that follows : chest X-ray, chest CT-scan and CT-angiography, bronchoscopy, ventilation-perfusion with single-photon emission computed tomography and pulmonary angiography in the diagnosis of different etiologies of hemoptysis.
All-cause mortality at 2 years | 2 years
  All-cause mortality at 2 years after the diagnosis of hemoptysis.
Smoking status | Day 1
  Determining the percentage of patients who : never smoked, is an active smoker, former smoker or unknown status.
Age | Day 1
  Determining the average age of the enrolled patients.
Gender | Day 1
  Determining the percentage of each gender of the enrolled patients.
International Normalized Ratio | Day 1
  Determining the median of the international normalized ratio (INR).
Partial Thromboplastin Time | Day 1
  Determining the median of the partial thromboplastin time (PTT).
Platelet count | Day 1
  Determining the average of the platelet count measured per microliter of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Grodin-Beaudoin, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hirshberg B, Biran I, Glazer M, Kramer MR. Hemoptysis: etiology, evaluation, and outcome in a tertiary referral hospital. Chest. 1997 Aug;112(2):440-4. doi: 10.1378/chest.112.2.440. PMID 9266882
- [Background] Jeudy J, Khan AR, Mohammed TL, Amorosa JK, Brown K, Dyer DS, Gurney JW, MacMahon H, Saleh AG, Vydareny KH; Expert Panel on Thoracic Imaging. ACR Appropriateness Criteria hemoptysis. J Thorac Imaging. 2010 Aug;25(3):W67-9. doi: 10.1097/RTI.0b013e3181e35b0c. PMID 20711032
- [Background] Alaoui AY, Bartal M, el Boutahiri A, Bouayad Z, Bahlaoui A, el Meziane A, Naciri A. [Clinical characteristics and etiology in hemoptysis in a pneumology service. 291 cases]. Rev Mal Respir. 1992;9(3):295-300. French. PMID 1615202
- [Background] Reechaipichitkul W, Latong S. Etiology and treatment outcomes of massive hemoptysis. Southeast Asian J Trop Med Public Health. 2005 Mar;36(2):474-80. PMID 15916059
- [Background] Sanai Raggad S, Abid H, Ghedira H, Tritar F, Hamzaoui A. [Current etiologies of hemoptysis in the elderly: comparative study of 360 cases]. Tunis Med. 2010 Nov;88(11):809-13. French. PMID 21049410
- [Background] Unsal E, Koksal D, Cimen F, Taci Hoca N, Sipit T. Analysis of patients with hemoptysis in a reference hospital for chest diseases. Tuberk Toraks. 2006;54(1):34-42. PMID 16615016
- [Background] Prasad R, Garg R, Singhal S, Srivastava P. Lessons from patients with hemoptysis attending a chest clinic in India. Ann Thorac Med. 2009 Jan;4(1):10-2. doi: 10.4103/1817-1737.43062. PMID 19561915
- [Background] Soares Pires F, Teixeira N, Coelho F, Damas C. Hemoptysis--etiology, evaluation and treatment in a university hospital. Rev Port Pneumol. 2011 Jan-Feb;17(1):7-14. doi: 10.1016/s2173-5115(11)70004-5. English, Portuguese. PMID 21251478
- [Background] Pedrol E, Fernandez-Sola J, Ferrer M, Barcelo J, Bosch X, Sande L, Camp J, Borras A, Urbano-Marquez A. [Hemoptysis: a prospective study of 108 cases in an emergency service]. Rev Clin Esp. 1991 May;188(9):450-4. Spanish. PMID 1896592
- [Background] Tsoumakidou M, Chrysofakis G, Tsiligianni I, Maltezakis G, Siafakas NM, Tzanakis N. A prospective analysis of 184 hemoptysis cases: diagnostic impact of chest X-ray, computed tomography, bronchoscopy. Respiration. 2006;73(6):808-14. doi: 10.1159/000091189. Epub 2006 Jan 27. PMID 16446530
- [Background] Wong CM, Lim KH, Liam CK. The causes of haemoptysis in malaysian patients aged over 60 and the diagnostic yield of different investigations. Respirology. 2003 Mar;8(1):65-8. doi: 10.1046/j.1440-1843.2003.00437.x. PMID 12856744
- [Background] Haro Estarriol M, Vizcaya Sanchez M, Jimenez Lopez J, Tornero Molina A. [Etiology of hemoptysis: Prospective analysis of 752 cases]. Rev Clin Esp. 2001 Dec;201(12):696-700. doi: 10.1016/s0014-2565(01)70953-8. Spanish. PMID 11835879